CLINICAL TRIAL: NCT04036136
Title: Development of a Novel Transdiagnostic Intervention for Anhedonia - R33 Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-2268b; R61MH110027 (NIH)
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2023-10

CONDITIONS: Anhedonia
MeSH Terms: conditions — Anhedonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation (Experimental): Treatment will consist of 15 weekly 45-minute sessions. Session 1 provides orientation and psychoeducation on anhedonia, and activity monitoring is introduced. Sessions 2-3 include structured values assessments of 10 life areas to enhance motivation for sustained behavior change and to clarify goals. Following goals clarification, an activity hierarchy is developed, establishing a set of idiographic behavioral targets across life areas prioritized by ease of implementation to scaffold task engagement during the course of treatment.
  Interventions: Behavioral: Behavioral Activation
- Mindfulness Treatment (Active Comparator): BATA will be compared to mindfulness based cognitive therapy (MBCT), chosen because its mechanisms of action are hypothesized to impact different brain mechanisms than BATA. Mindfulness is nonjudgmentally bringing awareness and acceptance to one's present-moment experience. MBCT will be administered in an individual format. The MBCT protocol will be modeled on the session outlines presented in Wahbeh et al., 2014. Treatment will be compromised of 15 weekly 45-minute sessions.
  Interventions: Behavioral: Mindfulness Treatment

INTERVENTIONS:
Behavioral: Behavioral Activation — Treatment will consist of 15 weekly 45-minute sessions.
  Arms: Behavioral Activation
Behavioral: Mindfulness Treatment — Treatment will consist of 15 weekly 45-minute sessions.
  Arms: Mindfulness Treatment

SUMMARY:
The overall goal of this project is to develop a novel transdiagnostic treatment for anhedonia, called Behavioral Activation Treatment for Anhedonia (BATA), using ultra-high field functional neuroimaging. There is a critical need for a validated treatment that specifically targets anhedonia, and this project will evaluate the effects of this new treatment on anhedonia and will establish how this treatment impacts brain systems that mediate reward processing, clinical symptoms of anhedonia, functional outcomes, and behavioral indices of reward processing. This work will also identify brain targets by which future novel anhedonia treatment may be evaluated.

DETAILED DESCRIPTION:
Deficits in motivation and pleasure, together referred to as anhedonia, are implicated in a number of psychiatric illnesses, including mood and anxiety disorders, substance-use disorders, schizophrenia, and attention-deficit/hyperactivity disorder. As a result, constructs related to anhedonia are central to the NIMH Research Domain Criteria (RDoC) project. Anhedonia is often one of the most difficult psychiatric symptoms to treat and thus represents a critical endophenotype and vulnerability factor for a range of psychiatric disorders. Given the centrality of anhedonia to a large number of psychiatric disorders, improved interventions to treat motivation and pleasure are critical for these disorders. The overall goal of this R61/R33 project is to develop a novel transdiagnostic treatment for anhedonia, called Behavioral Activation Treatment for Anhedonia (BATA). This new intervention is designed to treat anhedonia by emphasizing supported engagement with personally relevant goals and reducing avoidance behaviors. Consistent with the objectives and milestones outlined in RFA-MH-16-406 ("Exploratory Clinical Trials of Novel Interventions for Mental Disorders"), in the R61 phase of this trial that lasted from June 22, 2017-July 31, 2019, the investigators proposed to use an experimental therapeutics approach to first evaluate mesocorticolimbic target engagement by this treatment in a transdiagnostic sample characterized by clinically impairing anhedonia (Aim 1). Specifically, the investigators examined the effects of this treatment, relative to an active comparison treatment, on caudate nucleus activation during reward anticipation and rostral anterior cingulate cortex activation during reward outcomes using ultra-high field (7T) functional magnetic resonance imaging. The investigators also used fMRI to determine the optimal dose of the intervention (Aim 2).

In the current R33 phase of the study, which begins recruitment 8/1/2019, the investigators plan to evaluate the effects of the optimal dose of this new treatment, versus an active comparison treatment, on anhedonic symptoms and functional outcomes (Aim 3), behavioral indicators of reward sensitivity (Aim 4), and neural indicators of reward processing (Aim 5).

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old and treatment seeking;
* SHAPS scores ≥ 20, corresponding to clinically significant anhedonia;
* Clinician's Global Impression Scale-Severity score (CGI-S) > 3 to assure a clinically impaired sample;
* Seeking treatment for anhedonia (i.e., referred from an outpatient clinic or responded to an advertisement for anhedonia treatment; endorses desire for treatment during screening).

Exclusion Criteria:

* Those for whom medication management is the primary gold-standard treatment, including those with bipolar disorder/mania, schizophrenia spectrum, and other psychotic disorders;
* Prior treatment with behavioral activation therapy for depression or mindfulness-based treatments (those with exposure to other forms of psychotherapy, e.g., supportive therapy, will be eligible);
* Those who may have difficulty understanding the cognitive components of BATA, including those with intellectual disability, neurocognitive disorders, and dissociative disorders;
* Feeding and eating disorders which may have confounding effects on the fMRI signal;
* Substance Use Disorders given confounding effects of substances of abuse on the fMRI signal;
* Suicidal intent and plan;
* Psychotropic medication use in the past 4 weeks (8 weeks for fluoxetine) and/or current psychotherapy. Participants must be medication-free at study entry; study personnel will not supervise medication taper for the purpose of the study, but those who taper under the supervision of their regular provider will be eligible;
* Currently pregnant, as measured by urine pregnancy screen immediately before MRI scans;
* Positive urinalysis screen for cocaine, marijuana, opiates, methadone, amphetamines, and benzodiazepines (conducted on-site via Biosite Triage Meter Plus) at study entry.
* No neurological conditions (e.g., history of stroke, seizure, or TBI); Contraindications for fMRI imaging: Metal in the body, dental work that is not fillings or gold, any tattoos, any metal in the body, any metal injury - especially those to the eyes, any other type of implant unless they are 100% plastic.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel S Dichter, PhD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- UNC-Chapel Hill School of Medicine, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share de-identified data through the National Database for Clinical Trials Related to Mental Illness (NDCT)

REFERENCES:
- [Derived] Cernasov PM, Walsh EC, Nagy GA, Kinard JL, Kelley L, Phillips RD, Pisoni A, Diehl J, Haworth K, West J, Freeman L, Pfister C, Scott M, Daughters SB, Gaylord S, Dichter GS, Smoski MJ. A parallel-arm, randomized trial of Behavioral Activation Therapy for anhedonia versus mindfulness-based cognitive therapy for adults with anhedonia. Behav Res Ther. 2024 Nov;182:104620. doi: 10.1016/j.brat.2024.104620. Epub 2024 Aug 23. PMID 39213738
- [Derived] Gibson K, Cernasov P, Styner M, Walsh EC, Kinard JL, Kelley L, Bizzell J, Phillips R, Pfister C, Scott M, Freeman L, Pisoni A, Nagy GA, Oliver JA, Smoski MJ, Dichter GS. The effects of psychotherapy for anhedonia on subcortical brain volumes measured with ultra-high field MRI. J Affect Disord. 2024 Sep 15;361:128-138. doi: 10.1016/j.jad.2024.05.140. Epub 2024 May 28. PMID 38815760
- [Derived] Cernasov PM, Kinard JL, Walsh E, Kelley L, Phillips R, Pisoni A, Arnold M, Lowery SC, Ammirato M, Nagy GA, Oliver JA, Haworth K, Daughters SB, Dichter GS, Smoski M. Parsing within & between-person dynamics of therapy homework completion and clinical symptoms in two cognitive behavioral treatments for adults with anhedonia. Behav Res Ther. 2023 Jul;166:104322. doi: 10.1016/j.brat.2023.104322. Epub 2023 Apr 26. PMID 37148652
- [Derived] Phillips R, Walsh E, Jensen T, Nagy G, Kinard J, Cernasov P, Smoski M, Dichter G. Longitudinal associations between perceived stress and anhedonia during psychotherapy. J Affect Disord. 2023 Jun 1;330:206-213. doi: 10.1016/j.jad.2023.03.011. Epub 2023 Mar 11. PMID 36907457

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Activation: Treatment will consist of 8-15 weekly 45-minute sessions. Session 1 provides orientation and psychoeducation on anhedonia, and activity monitoring is introduced. Sessions 2-3 include structured values assessments of 10 life areas to enhance motivation for sustained behavior change and to clarify goals. Following goals clarification, an activity hierarchy is developed, establishing a set of idiographic behavioral targets across life areas prioritized by ease of implementation to scaffold task engagement during the course of treatment.
  Behavioral Activation: Treatment will consist of 8-15 weekly 45-minute sessions.
- Mindfulness Treatment: Behavioral Activation Therapy for Anhedonia (BATA) will be compared to mindfulness based cognitive therapy (MBCT), chosen because its mechanisms of action are hypothesized to impact different brain mechanisms than BATA. Mindfulness is nonjudgmentally bringing awareness and acceptance to one's present-moment experience. MBCT will be administered in an individual format. Treatment will be compromised of 8-15 weekly 45-minute sessions.
  Mindfulness Treatment: Treatment will consist of 8-15 weekly 45-minute sessions.
Period: Overall Study
Arm/Group | Behavioral Activation | Mindfulness Treatment
Started | 61 | 55
Completed | 46 | 35
Not Completed | 15 | 20

BASELINE CHARACTERISTICS:
Groups:
- Mindfulness Treatment: BATA will be compared to mindfulness based cognitive therapy (MBCT), chosen because its mechanisms of action are hypothesized to impact different brain mechanisms than BATA. Mindfulness is nonjudgmentally bringing awareness and acceptance to one's present-moment experience. MBCT will be administered in an individual format. The MBCT protocol will be modeled on the session outlines presented in Wahbeh et al., 2014. Treatment will be compromised of 8-15 weekly 45-minute sessions.
  Mindfulness Treatment: Treatment will consist of 8-15 weekly 45-minute sessions.
- Total: Total of all reporting groups
Arm/Group | Behavioral Activation | Mindfulness Treatment | Total
Number analyzed (Participants) | 61 | 55 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.26 (8.51) | 30.20 (9.45) | 29.18 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 79
  Male | 20 | 17 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 56 | 45 | 101
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 14 | 9 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 31 | 34 | 65
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 55 | 116

OUTCOME MEASURES:

1. Primary Outcome: Change in Snaith-Hamilton Pleasure Scale Score Over Time
Description: The Snaith-Hamilton Pleasure Scale (SHAPS), a well-validated 14-item questionnaire will be used to assess hedonic capacity. The sum of the 14 items scores ranges from 0 to 56. A higher score represents more anhedonic symptoms. Treatment duration varied across participants. Participants participated in as few as 8 weekly sessions or in as many as 15 weekly sessions of psychotherapy, based on therapist judgement. Thus the outcome measure timeframe varied between 8 and 15 weeks.
Time Frame: Baseline, Post-treatment (between 8 to 15 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation | Mindfulness Treatment
Number analyzed (Participants) | 61 | 55
score on a scale
  Baseline | 37.67 (3.73) | 36.96 (4.75)
  Last observation (up to Week 15) | 29.62 (5.15) | 29.76 (6.90)
Statistical Analysis 1: Comparison: Behavioral Activation vs Mindfulness Treatment; Model covariates are Baseline SHAPS, age, and sex; Test type: Equivalence — The equivalence margin is 0; p = 0.724, ANCOVA; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-2.41 to 1.68]

2. Secondary Outcome: Change in Neural Activation During MID Task Anticipation Phase
Description: Neural activation assessed by Functional Magnetic Resonance Imaging (fMRI) during Monetary Incentive Delay (MID) task. During MID the task, participants respond to "win" trials by pressing a button on a button box in the MRI as quickly as possible when the see a target. MID task reward anticipation is defined by the contrast in fMRI signal between reward and neutral trials during the presentation of cues and the fixation cross. Because this subtraction method is used to define the fMRI signal, it is possible for this value to be negative. Treatment duration varied across participants. Participants participated in as few as 8 weekly sessions or in as many as 15 weekly sessions of psychotherapy, based on therapist judgement. Thus the outcome measure timeframe varied between 8 and 15 weeks.
Time Frame: Baseline, Post-treatment (between 8 to 15 weeks)
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Behavioral Activation | Mindfulness Treatment
Number analyzed (Participants) | 47 | 39
percent signal change
  Baseline | -0.030 (0.172) | 0.052 (0.162)
  Last observation (up to Week 15) | -0.001 (0.176) | 0.046 (0.182)
Statistical Analysis 1: Comparison: Behavioral Activation vs Mindfulness Treatment; Model covariates are Baseline fMRI, age, and sex; Test type: Equivalence — The equivalence margin is 0; p = 0.292, Regression, Linear; Mean Difference (Final Values) = -0.043, 95% CI 2-sided [-0.124 to 0.038]

3. Secondary Outcome: Change in Neural Activation During MID Task Outcome Phase
Description: Brain activation assessed by Functional Magnetic Resonance Imaging (fMRI) during Monetary Incentive Delay (MID) task. During MID the task, participants respond to "win" trials by pressing a button on a button box in the MRI as quickly as possible when the see a target. MID task reward outcome is defined by the contrast in fMRI signal between successful and unsuccessful reward trials during the presentation of feedback. Because this subtraction method is used to define the fMRI signal, it is possible for this value to be negative.
Time Frame: up to 15 weeks
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Behavioral Activation | Mindfulness Treatment
Number analyzed (Participants) | 47 | 39
percent signal change
  Baseline | 0.349 (0.416) | 0.271 (0.387)
  Last observation (up to Week 15) | 0.114 (0.374) | 0.263 (0.371)
Statistical Analysis 1: Comparison: Behavioral Activation vs Mindfulness Treatment; Model covariates are Baseline fMRI, age, and sex; Test type: Equivalence — The equivalence margin is 0; p = 0.084, Regression, Linear — The equivalence margin is 0; Median Difference (Final Values) = -0.148, 95% CI 2-sided [-0.316 to 0.020]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of signing informed consent through final MRI sessions. Due to the design of the trial, each participant was in the trial for between 8-15 weeks.
Arm/Group | Behavioral Activation | Mindfulness Treatment
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/55
Other Adverse Events (participants affected / at risk) | 4/61 | 11/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Activation (N=61) | Mindfulness Treatment (N=55)
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT04036136/Prot_SAP_000.pdf